CLINICAL TRIAL: NCT01132001
Title: EVALUATION OF BLOOD PRESSURE MEASUREMENTS OUTSIDE OFFICE: COMPARISON OF DIAGNOSIS BASED ON EITHER AMBULATORY OR HOME BLOOD PRESSURE MEASUREMENTS
Brief Title: Ambulatory Versus Home Blood Pressure Measurement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Other Study IDs: HBP5
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective study comparing the three blood pressure monitoring methods on the diagnosis of arterial hypertension. Blood pressure of each subject will be evaluated with clinic, home and 24h ambulatory blood pressure measurements in three visits

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 yrs
* Patients referred to an outpatient clinic for high blood pressure
* Patients with no treatment or with antihypertensive treatment stable for at least 4 weeks.
* Patients capable of performing home blood pressure measurements.
* Signed informed consent

Exclusion Criteria:

* Hypertension stage III (SBP>180 mmHg or DBP>110mmHg)
* Secondary hypertension
* Resistant hypertension
* Arrhythmia
* Pregnancy
* Symptomatic heart disease
* Renal disease (Cr>2mg/dl)
* Uncontrolled diabetes mellitus (HbA1c>8.5%)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred to an outpatient hyperetension clinic for arterial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure monitoring methods | Baseline
  Comparison among clinic, home and ambulatory blood pressure measurements.

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, MD, Study Chair — Hypertension Center,Third Department of Medicine,University of Athens,Greece
Locations (1):
- Hypertension Center, Third Department of Medicine, University of Athens, Greece, Athens, Greece